CLINICAL TRIAL: NCT01734096
Title: Effect of Lower Body Negative Pressure and Angiotensin II Receptor Blockade on Renal Hemodynamic, Neuro-hormonal and Tubular Response in Pre-hypertensive States: a Randomized Controlled Trial.
Brief Title: Renal Response to Lower Body Negative Pressure in Pre-hypertensive States
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PD Dr. Grégoire Wuerzner (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, PD Dr. Grégoire Wuerzner, Doctord, MD, privat docent, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PZ00P3_121655
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Hypertension; Obesity; White Coat Hypertension; Resistant Hypertension
Keywords: hypertension; obesity; white coat hypertension; resistant hypertension
MeSH Terms: conditions — Hypertension; Obesity; White Coat Hypertension | interventions — Lower Body Negative Pressure; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- control group (Active Comparator): healthy volunteer
  Interventions: Other: Lower body negative pressure (LBNP); Drug: Candesartan cilexetil
- obesity group (Active Comparator): Patients with BMI >30 Kg/m2
  Interventions: Other: Lower body negative pressure (LBNP); Drug: Candesartan cilexetil
- white coat hypertension group (Active Comparator): Patients with office blood pressure >140/90 mmHg and ambulatory daytime blood pressure <135/85 mmHg
  Interventions: Other: Lower body negative pressure (LBNP); Drug: Candesartan cilexetil
- Resistant hypertension (Active Comparator): Patients with ambulatory blood pressure > 135/85 mm Hg (day) or >120/70 mm Hg (night) with 3 antihypertensive drugs with direct observance of drug taking.
  Interventions: Other: Lower body negative pressure (LBNP)

INTERVENTIONS:
Other: Lower body negative pressure (LBNP) — Lower limbs are put in in LBNP device for one hour (-30 mbar)
Drug: Candesartan cilexetil — candesartan cilexetil 16 mg once a day for 7 days cross over with placebo in control group, obesisty group and white coat hypertension group
  Arms: control group; obesity group; white coat hypertension group

SUMMARY:
The purpose of this study is to determine whether in pre-hypertensive and hypertensive states such as white coat hypertension, obesity related hypertension or resistant hypertension, renal function is more sensitive to orthostatic stress.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 Kg/m2 (obesity group)
* office BP >140/90 and daytime ambulatory blood pressure <135/85 (white coat hypertension group) _daytime abpm >135/85 mm Hg or nighttime abpm 120/70

Exclusion Criteria:

* History of allergic reaction
* Diabetes type 1 or type 2
* History of renal artery stenosis
* Acute illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-05; Primary Completion 2013-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
sodium excretion | after one hour of lower body negative pressure
  sodium excretion will be compared to control group (healthy volunteers) after one hour of lower negative pressure. The protocol includes 2 hours of baseline measure, one hour of lower negative pressure and 2 hours of recovery

SECONDARY OUTCOMES:
glomerular filtration rate | after one hour of lower body negative pressure

OTHER OUTCOMES:
renal plasma flow | after one hour of lower body negative pressure

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire Wuerzner, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Michel Burnier, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Switzerland (2):
  - Service of nephrology and hypertension, Lausanne, Canton of Vaud
  - Service of nephrology and hypertension, Lausanne

REFERENCES:
- [Derived] Vakilzadeh N, Petrovic D, Maillard M, Favre L, Grouzmann E, Wuerzner G. Impact of obesity with or without hypertension on systemic haemodynamic and renal responses to lower body negative pressure. Blood Press. 2021 Feb;30(1):67-74. doi: 10.1080/08037051.2020.1829963. Epub 2020 Oct 19. PMID 33073631
- [Derived] Vuignier Y, Grouzmann E, Muller O, Vakilzadeh N, Faouzi M, Maillard MP, Qanadli SD, Burnier M, Wuerzner G. Blood Pressure and Renal Responses to Orthostatic Stress Before and After Radiofrequency Renal Denervation in Patients with Resistant Hypertension. Front Cardiovasc Med. 2018 May 23;5:42. doi: 10.3389/fcvm.2018.00042. eCollection 2018. PMID 29876358